CLINICAL TRIAL: NCT04526132
Title: A Multi-center, Randomized, Double-blind, Placebo Parallel Controlled Phase Ⅲ Clinical Trial on the Efficacy and Safety of Felbinac Trometamol Injection in the Treatment of Moderate and Severe Postoperative Pain
Brief Title: A Phase Ⅲ Clinical Study Trial of Felbinac Trometamol Injection in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BALF-PAIN-3001
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: group1 (Experimental): Generic name: Felbinac Trometamol Injection; Placebo:Normal saline Dosage form: Injection Dosage:8ml Volume:4ml
  Interventions: Drug: Felbinac Trometamol Injection
- Experimental: group2 (Placebo Comparator): Generic name:Placebo Placebo:Normal saline Dosage form:Injection Dosage:8mg Volume:4ml
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Felbinac Trometamol Injection — Felbinac Trometamol Injection diluted to 100 ml with 0.9% sodium chloride injection.Use a micro-injection pump to inject intravenously at a constant speed for 30 min (± 2 min)..
  One dose at 8h、16h 、24h、32h and 40h after the start of the first dose,the first intravenous infusion was started at the end of the operation (Skin suture completes the last stitch).The drug was given 6 times,3 times/day,once every 8 hours.
  Other Names: 4-Biphenylacetic Acid Trishydroxymettiylaminometnane
  Arms: Experimental: group1
Drug: Placebos — Placebo diluted to 100 ml with 0.9% sodium chloride injection.Use a micro-injection pump to inject intravenously at a constant speed for 30 min (± 2 min).
  One dose at 8h、16h 、24h、32h and 40h after the start of the first dose,the first intravenous infusion was started at the end of the operation (Skin suture completes the last stitch).The drug was given 6 times,3 times/day,once every 8 hours.
  Other Names: Normal saline
  Arms: Experimental: group2

SUMMARY:
A multi-center, randomized, double-blind, placebo parallel controlled phase Ⅲ clinical trial on the efficacy and safety of felbinac trometamol Injection in the treatment of moderate and severe postoperative pain.main purpose is to evaluate the efficacy of Felbinac Trometamol Injection in the treatment of moderate and severe pain after surgery.Secondary purpose is to evaluation the safety of Felbinac Trometamol Injection in the treatment of moderate and severe pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18≤age≤65 years of age, gender is not limited;
* ASA grade I or II;
* 18 ≤ body mass index (BMI) ≤ 30 [BMI = weight (kg) / height 2 (m2)];
* Expected hospital stay ≥72 hours after surgery；
* Patients planned to receive laparotomy or laparoscopic upper abdominal surgery with a single surgical incision ≥5 cm, thoracoscopic chest surgery (such as lung lobe resection surgery, lung wedge resection surgery, etc.),both under general anesthesia;
* Expected to require more than 48 hours of PCIA (patient controlled intravenous analgesia) treatment after surgery;
* Ability to understand research procedures and pain scales, operate PCIA devices, and communicate effectively with researchers;
* Agree to participate in the trial and voluntarily sign the informed consent form.

Exclusion Criteria:

* Except for the chronic pain caused by the target lesion of this operation, those who have a history of chronic pain for more than 3 months or who are undergoing regular analgesia for more than 3 months;
* Those who have used barbiturates within 20 days before surgery, those who used other analgesics, muscle relaxants or sedatives within 24 hours before operation (excluding those required for this operation), or those who used long-acting non-steroidal anti-inflammatory drugs (NSAIDs) within 12 hours, or those who used short-acting non-steroidal anti-inflammatory drugs (NSAIDs) within 6 hours before operation.
* A person with high bleeding risk, and also including who with congenital bleeding disorders (such as hemophilia), thrombocytopenia (PLT < 80 × 10 ∧ 9 / L), abnormal platelet function (such as idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital platelet dysfunction, etc.) or any clinically significant active bleeding, coagulopathy;
* A person who received full-dose anticoagulant therapy, activated protein C or thrombolytic drugs within 6 hours before surgery (except for heparin subcutaneous injection for preventive treatment);
* People with heart failure (NYHA grade III or IV), unstable angina pectoris, acute myocardial infarction, and severe arrhythmia within 6 months before surgery
* Hypertensive patients who have not been satisfactorily controlled by blood pressure (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥105mmHg), or ACEI/diuretics for ≥30 days, or hypotension (systolic blood pressure <90mmHg);
* People with pulmonary heart disease or other serious respiratory diseases that are not the purpose of this treatment;
* Person with gastrointestinal ulcer and a history of gastrointestinal bleeding 6 months before operation and required medical treatment(prophylactic medication or undiagnosed persons are not excluded);
* Those with previous cerebral arteriovenous malformations, cerebral aneurysms, brain tumors, or preoperative traumatic brain injury, intracranial surgery, history of stroke;
* Patients with poor glycemic control of diabetes (random blood glucose > 11.1mmol / L);
* Patients with autoimmune diseases, connective tissue diseases, etc. who need long-term use of adrenocortical hormone therapy;
* Abnormal liver and kidney function: ALT/AST> 2 times the upper limit of normal value, or creatinine> upper limit of normal value, or dialysis treatment within 28 days before surgery;
* Allergic constitution, or known to be allergic to this drug, NSAIDs, and opioids;
* Patients who are afflicted with narcotic drugs, drugs, or resistant to opioids;
* A woman who is breast-feeding or pregnant, who is unable or unwilling to follow the investigator's guidance during the study period and within 3 months after the last study treatment;
* Those who have participated in other clinical trials within 3 months before surgery;
* Investigators believe that it is not suitable for participating in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
24h total morphine consumption | up to 24hours after multi-dose
  The total amount of morphine within 24 hours after the end of first drug administration

SECONDARY OUTCOMES:
Area under the pain intensity curve during movement (AUCM) | 0-8 h，8-16 h，16-24 h and 0-48 h
  Pain intensity under movement
Area under the pain intensity curve during rest(AUCR) | 0-8 h，8-16 h，16-24 h and 0-48 h
  Pain intensity under rest
Pain intensity at 48 hours after the end of the first administration under movement | up to 48 hours after multi-dose
Pain intensity at 48 hours after the end of the first administration under rest | up to 48 hours after multi-dose
Press time | up to 48 hours after multi-dose
  The first time to press the analgesic pump for analgesia
Total and effective pressing times of analgesic pump | up to 24 and 48 hours after multi-dose
The proportion of morphine used to remedy analgesia | up to 24 and 48 hours after multi-dose
Total amount of morphine administered within 48 hours after the first administration | up to 48 hours after multi-dose

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ouyang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- Shijiazhuang Yiling Pharmaceutical Co.,Ltd, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No